CLINICAL TRIAL: NCT01578811
Title: Study to Assess the Efficacy and Safety of SK-MS10 in Subjects With Acute and Chronic Gastritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SK-MS10_GID_II_2010
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2010-12

CONDITIONS: Erosive Gastritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- SK-MS10 160mg t.i.d (Experimental)
  Interventions: Drug: SK-MS10
- SK-MS10 320mg t.i.d (Experimental)
  Interventions: Drug: SK-MS10

INTERVENTIONS:
Drug: Placebo — Dosage
  Arms: Placebo
Drug: SK-MS10 — Dosage
  Arms: SK-MS10 160mg t.i.d
Drug: SK-MS10 — Dosage
  Arms: SK-MS10 320mg t.i.d

SUMMARY:
The purpose of this study is to Assess the Efficacy and Safety of SK-MS10 in subjects With acute and chronic gastritis.

ELIGIBILITY:
Inclusion Criteria:

1. Have been diagnosed as erosive gastritis by endoscopy within 1 weeks before enrollment.
2. Patients who voluntarily signed written informed consent may participate in the study.

Exclusion Criteria:

1. Pregnant or lactating female.
2. Patients have gastric ulcer, duodenal ulcer and GERD.
3. Use of any proton pump inhibitor, H2-receptor antagonist, muscarine receptor antagonist and gastrin receptor antagonist within 2 weeks before initiating study drug therapy
4. Patients requiring corticosteroid therapy
5. Severe neurological or psychological disease
6. History of allergic reaction to the medications used in this study
7. Use of other investigational drugs within 30 days prior to the study.
8. Patients that investigators consider ineligible for this study

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improvement rates of erosive gastritis according to the sydney classification | Change from Baseline in the grade of erosive gastritis at 2 weeks

SECONDARY OUTCOMES:
Healing rates of erosive gastritis according to the sydney classification | Change from Baseline in the grade of gastric erosions at 2 weeks
Improvement rates of erosive gastritis by estimated the number of erosion | Change from Baseline in the number of gastric erosions at 2 weeks
Healing rates of edema according to the sydney classification | Change from Baseline in the grade of edema at 2 weeks
Improvement rates of erythema according to the sydney classification | Change from Baseline in the grade of erythema at 2 weeks
Improvement rates of hemorrhage according to the Scandinavian Journal of Gastroenterology - Supplement | Change from Baseline in the grade of hemorrhage at 2 weeks
Improvement rates of symptoms using Korean NDI | Questionaire at baseline and then week 2

CONTACTS AND LOCATIONS:
Locations (1):
- SKChemicals, Seoul, South Korea